CLINICAL TRIAL: NCT06836726
Title: Phase II Clinical Trial to Test Efficacy of Targeting Hypoxia Combined With ARSI After First-line ARSI Therapy for Castrate Resistant Prostate Cancer
Brief Title: Clinical Trial to Test Efficacy of Targeting Hypoxia Combined With ARSI After First-line ARSI Therapy for Castrate Resistant Prostate Cancer
Acronym: EVO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: ImmunoGenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-6044
Record Dates: First submitted 2025-02-03; First posted 2025-02-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: CRPC; Castration Resistant Prostate Cancer; ARSIs; androgen receptor signal inhibitors
MeSH Terms: interventions — TH 302

STUDY DESIGN:
Intervention Model Description: This is a single-institution, single-arm, open-label Phase 2 trial evaluating evofosfamide in subjects with M1 CRPC who fail first-line ARSIs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluating evofosfamide in subjects with M1 CRPC who fail first-line ARSIs (Experimental): After baseline molecular imaging (PSMA and fluorodeoxyglucose (FDG) PET/CT), prior to evofosfamide initiation, subjects will be encouraged to undergo biopsy of a dominant lesion: FDG-, PSMA-uptake and/or conventional imaging determined (in order, and according to feasibility). Subjects will then receive the alternate ARSI (i.e., different from the one received in first line) as per current standard practice and Provincial drug plan coverage. Additionally, subjects will receive combinatorial evofosfamide at a dose of 480 mg/m2 intravenously (IV) over 60 minutes on Days 1, 8 and 15 of every 28-day cycle. Therapy will continue until disease progression, unacceptable toxicity as a result of evofosfamide, or subject withdrawal. Assessments during evofosfamide treatment will include history, physical exam, and blood tests at each monthly visit to monitor for toxicity. Subjects will be followed for survival endpoints following completion of this study treatment until death.
  Interventions: Drug: Evofosfamide

INTERVENTIONS:
Drug: Evofosfamide — This study is evaluating evofosfamide in subjects with M1 CRPC who fail first-line ARSIs.

SUMMARY:
This is a single-institution, single-arm, open-label Phase 2 trial evaluating evofosfamide in subjects with M1 CRPC who fail first-line ARSIs. In those progressing after second-line Docetaxel or deemed ineligible to it, the use of alternate ARSI remains the most common line of therapy in our Province, in keeping with recent international recommendations. After baseline molecular imaging (PSMA and fluorodeoxyglucose (FDG) PET/CT), prior to evofosfamide initiation, subjects will be encouraged to undergo biopsy of a dominant lesion: FDG-, PSMA-uptake and/or conventional imaging determined (in order, and according to feasibility). Subjects will then receive the alternate ARSI (i.e., different from the one received in first line) as per current standard practice and Provincial drug plan coverage. Additionally, subjects will receive combinatorial evofosfamide at a dose of 480 mg/m2 intravenously (IV) over 60 minutes on Days 1, 8 and 15 of every 28-day cycle. Therapy will continue until disease progression, unacceptable toxicity as a result of evofosfamide, or subject withdrawal. Assessments during evofosfamide treatment will include history, physical exam, and blood tests at each monthly visit to monitor for toxicity. Response and progression will be evaluated by whole-body PSMA PET/CT scan every 8 weeks (± 3 days) and determined using (PE)RECIST v1.1 criteria. PSA, NE markers (e.g., Serum CHGA, NSE), organ function tests (e.g., liver, kidney) and investigational liquid biopsy samples will be followed every cycle (monthly). FDG PET/CT will be performed at baseline, at 6-10 weeks from the date of signing the informed consent form (ICF), and upon progression, irrespective of treatment discontinuation or initiation of another therapy. Subjects will be followed for survival endpoints following completion of this study treatment until death.

DETAILED DESCRIPTION:
Evofosfamide at a dose of 480 mg/m2 IV over 60 minutes on Days 1, 8 and 15 of every 28-day cycle. Additionally, subjects will receive standard-of-care castration (medical or surgical) plus ARSI. On days when both an ARSI and evofosfamide are administered, the ARSI should be administered at least 2 hours before or at least 2 hours after completion of the evofosfamide infusion. The preferred order of administration is evofosfamide administered first, with the ARSI administered at least 2 hours following the completion of evofosfamide infusion.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age;
2. Ability to understand the purposes and risks of the trial and has signed a written ICF approved by the investigator's REB;
3. CRPC stage M1 based on conventional imaging (CT and/or bone scan) or PSMA PET;
4. Progression (i.e., PSA rise of 25% or more, and absolute increase of 2 ng/mL or more from the nadir) to first-line ARSIs (Abi or Enza or Daro or Apa monotherapy) and subsequent docetaxel or deemed ineligible for it;
5. Ongoing castration therapy (e.g., surgical or medical with LHRH agonists/antagonist), with baseline testosterone level <50ng/dL;
6. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2;
7. In subjects with known significant pulmonary disease (severe chronic obstructive or other pulmonary disease with hypoxemia), measure oxygen saturation using pulse oximeter after a 2-minute walk. Subjects must have oxygen saturation ≥90% to be eligible for the trial.

Exclusion Criteria:

* 1. ANC <1,000/mm3, and/or hemoglobin <9.0 g/dL, and/or platelet count <100,000/mm3; independent of transfusion and/or growth factors 2. Liver dysfunction: total bilirubin, serum glutamic oxaloacetic transaminase (SGOT; aspartate aminotransferase [AST]) and/or serum glutamic-pyruvic transaminase (SGPT; alanine aminotransferase [ALT]) >1.5 × upper normal limit (UNL); 3. Inadequate renal function: creatinine >1.5 × UNL, or eGFR <40 mL/min; 4. Any Grade 3 or greater toxicity experienced during treatment with prior ARSI; 5. Severe, active co-morbidity defined as follows:

  1. Myocardial infarction within 6 months prior to date of enrollment.
  2. Current severe or unstable angina.
  3. New York Heart Association Functional Classification III/IV. (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
  4. Severe chronic obstructive or other pulmonary disease with hypoxemia at rest (requires supplementary oxygen, symptoms due to hypoxemia).
  5. History of any condition that in the opinion of the investigator, would preclude participation in this study.

     6. Known liver metastases based on conventional imaging (i.e., abdominal CT and/or MR).

     7. Known brain, leptomeningeal or epidural metastases (unless treated, well controlled, and not requiring steroidal therapy for at least 3 months).

     8. Major surgery (other than diagnostic surgery), open biopsy, or significant traumatic injury, ≤28 days prior to the date of signing informed consent. Subject must have completely recovered from surgery.

     9. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.

     10. Treatment of PCa with radiation therapy or surgery ≤28 days prior to the Cycle 1 Day 1.

     11. Prior therapy with a hypoxic cytotoxin. 12. HIV-infected patients with detectable viral load and/or on effective anti-retroviral therapy (ART) with undetectable viral load for less than 6 months. Note: HIV testing is not required for eligibility for this protocol. Drug-drug interactions with ART occur via many mechanisms, with cytochrome P450 CYP3A4-mediated interactions being the most common. Patients who are using concurrent strong or moderate CYP3A4 inhibitors (e.g., ritonavir, cobicistat) or strong or moderate CYP3A4 inducers must be switched to an alternate effective ART regimen ≥4 weeks before study enrollment or should be excluded from the study if their regimen cannot be altered.

     13. Active infection with hepatitis B or hepatitis C (i.e., detectable viral load) with or without active treatment in patients with previously known infection. Note: Only Hepatitis B testing is required for eligibility for this protocol as per standard practice prior to systemic therapy.

     14. Subjects who have exhibited allergic reactions to a structural compound similar to evofosfamide or the drug product excipients.

     15. Subjects who are taking medications that prolong QT interval and have a risk of Torsades de Pointes (see Appendix A).

     16. Subjects with a QTc interval calculated according to Fridericia formula (QTC = QT / RR1/3) of >450 msec based on screening electrocardiogram (ECG).

     17. Subjects with a history of long QT syndrome. 18. Subjects taking a medication that is a moderate or strong inhibitor or inducer of CYP3A4within 14 days or 5 half-lives (whichever is longer) prior to signing of ICF. (see Appendix B).

     19. Subjects taking a medication that is a sensitive substrate or substrates with a narrow therapeutic index of CYP3A4, CYP2D6, or CYP2C9 (see Appendix C).

     20. Any other significant concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this trial.

     21. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2026-05-27 (Estimated); Primary Completion 2028-05-27 (Estimated); Study Completion 2030-05-27 (Estimated)

PRIMARY OUTCOMES:
Preliminary clinical efficacy measures of evofosfamide in subjects with CRPC progressing to first-line ARSIs +/- docetaxel | Every 8 weeks (± 3 days) until death
  Preliminary clinical efficacy measures of evofosfamide in subjects with CRPC (Castrate Resistant Prostate Cancer) progressing to first-line ARSIs (Androgen Receptor Signaling Inhibitor) +/- docetaxel will be determined. This is measured by the biochemical response rate (if the PSA (tumor marker) declined ≥50% compared to baseline). Sample(s) may be drawn with serum biochemistry sample(s).

SECONDARY OUTCOMES:
Radiological (morphological and molecular) response rates | Every 8 weeks (± 3 days) until death
  Radiologic response rates (morphologic and molecular) measured using (PE)RECIST (Response evaluation criteria in solid tumors) criteria v1.1 on prostate-specific membrane antigen (PSMA) positron emission tomography (PET)/ computerized tomography (CT).
Professional free survival (PFS) | Every 8 weeks (± 3 days) until death
  PFS (progression free survival) from time of first evofosfamide treatment until biochemical [increase in PSA (tumor marker) >25% or an absolute increase of >2 ng/mL over baseline or nadir].
Response rate and PFS (progression free survival) to subsequent therapies (PFS2) | Every 8 weeks (± 3 days) until death
  Radiological or clinical progression; occurrence rate and time-to-event of NEPC phenotype based on histological (e.g., small cell NEPC or adenocarcinoma with >50% staining to CHGA and/or SYP and/or NSE), clinical (e.g., development of visceral metastases without biochemical progression) or biochemical (e.g., serum CHGA level >5× and/or NSE >2× UNL); response rate and PFS2.
OS (overall survival) | Every 8 weeks (± 3 days) until death
  OS (overall survival) as time from first treatment until death.
Changes in tumor biopsies | Every 8 weeks (± 3 days) until death
  Toxicity rates graded by CTCAE v5.0 (Common Terminology Criteria for Adverse Events).
Circulating cfDNA markers in response to therapy | Every 8 weeks (± 3 days) until death
  Circulating cfDNA markers will be determined in response to therapy via molecular analyses on pre- and during-treatment tissue and/or liquid biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada